CLINICAL TRIAL: NCT05537779
Title: Safety and Performance of Optivantage Multi-use Solution When Injecting Contrast Media to Subjects Requiring Contrast Enhanced CT Examination
Brief Title: Safety and Performance of Optivantage Multi-use When Injecting Contrast Media for Contrast Enhanced CT Examination
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: OPV-88-001
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Patient Participation
Keywords: Safety; Performance; Power Injector; Optivantage
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CT examination — Administration of contrast medium using the power injector

SUMMARY:
The study is a prospective, single-arm observational multicenter clinical investigation.

The primary objective is to confirm the safety and performance of the Optivantage® Injection System when injecting contrast media to subjects requiring contrast-enhanced CT imaging, in multi-patient use.

DETAILED DESCRIPTION:
Each subject will undergo CT examination in multi-use context using Optivantage Dual-head Contrast Delivery System.

100 subjects are expected to be enrolled. The safety and performance of the injector will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject referred for a contrast-enhanced CT examination using a power injector
* Subject or legal representative for children, having provided written informed consent

Exclusion Criteria:

* Subject weighting less than 10 kg
* Pregnant or breastfeading woman subject
* Subject with known allergy or hypersensitivity to contrast media
* Subject has contra-indication(s) to CT scanner and/or contrast medium as per the Summary of Product Characteristics
* Subject with peripherally inserted central catheter, central venous line, or port-A-catheter inserted for injection
* Subject unlikely to comply with the CIP, e.g. uncooperative attitude and unlikelihood of completing the study

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects referred for contrast enhanced CT examination who meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Safety of Optivantage | Per procedure
  Rate of extravasation
Performance of Optivantage | Per procedure
  Success of injection

SECONDARY OUTCOMES:
Safety of Optivantage | Per procedure
  Rate of patient complications
Device deficiencies | Per procedure
  Rate of device deficiencies including malfunction and error use